CLINICAL TRIAL: NCT01059097
Title: Effect of Surgeon Volume on Outcome of Pancreaticoduodenectomy in a High Volume Hospital.
Brief Title: Effect of Surgeon Volume on Outcome of Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Marco Braga, MD, San Raffaele University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANCREAS2010
Record Dates: First submitted 2010-01-25; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Cancer; Pancreatic Surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume surgeons (Active Comparator): high volume surgeons performed at least 18 PD/year.
  Interventions: Procedure: Pancreaticoduodenectomy
- Low volume surgeons (Active Comparator): low volume surgeons performed less than 18 PD/year.
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy

SUMMARY:
The independent impact of surgeon volume on outcome of patients undergoing pancreaticoduodenectomy in a high-volume Institution was assessed. A significant reduction of pancreatic fistula rate was found in the high-volume surgeon group in comparison with low-volume surgeon group. However, no difference between groups was found in mortality, major complications, and hospital stay.

DETAILED DESCRIPTION:
Objectives: To define the independent impact of surgeon volume on outcome after pancreaticoduodenectomy (PD) in a single high-volume institution.

Summary Background Data: The impact of surgeon volume on PD outcome is still controversial. So far, data available are from retrospective multi-institutional reviews, considering in-hospital mortality as the only outcome variable.

Methods: Prospectively collected data on 610 patients who underwent PD from August 2001 to August 2009 were analyzed. Cut-off value to categorize high and low-volume surgeons (HVS and LVS, respectively) was 18 PD/year. Primary endpoint was operative mortality (death within 30-day post-discharge). Secondary endpoints were morbidity, pancreatic fistula (PF) and length of stay. Demographic, clinical, and surgical variables were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreaticoduodenectomy between August 2001 and August 2009

Exclusion Criteria:

* Other type of surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2001-08; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality after pancreaticoduodenectomy within 30 days of discharge | 30 days after discharge

SECONDARY OUTCOMES:
Postoperative morbidity rate measuring the following complications: pancreatic fistula, biliary fistula, delayed gastric emptying, infectious complications, bleeding, cardiovascular complications, respiratory complications. | 30 days post-discharge
Postoperative hospital stay. Measuring the length of hospital stay. | At day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Principal Investigator — San Raffaele University
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy

REFERENCES:
- [Background] Balzano G, Zerbi A, Braga M, Rocchetti S, Beneduce AA, Di Carlo V. Fast-track recovery programme after pancreatico- duodenectomy reduces delayed gastric emptying. Br J Surg. 2008 Nov;95(11):1387-93. doi: 10.1002/bjs.6324. PMID 18844251
- [Background] Balzano G, Zerbi A, Capretti G, Rocchetti S, Capitanio V, Di Carlo V. Effect of hospital volume on outcome of pancreaticoduodenectomy in Italy. Br J Surg. 2008 Mar;95(3):357-62. doi: 10.1002/bjs.5982. PMID 17933001